CLINICAL TRIAL: NCT00001009
Title: A Phase I/II Dose Ranging Trial of Oral Dextran Sulfate (UA001) in HIV Infected Individuals and in Patients With Acquired Immunodeficiency Syndrome (AIDS) or AIDS Related Complex (ARC)
Brief Title: A Study of Dextran Sulfate in HIV-Infected Patients and in Patients With AIDS or AIDS Related Complex (ARC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: ACTG 060; 11034 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: T-Lymphocytes; HIV Antigens; Dextran Sulfate; Dose-Response Relationship, Drug; Drug Evaluation; Drug Therapy, Combination; Acquired Immunodeficiency Syndrome; AIDS-Related Complex
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Dextran Sulfate

INTERVENTIONS:
Drug: Dextran sulfate

SUMMARY:
To determine the effectiveness and safety of dextran sulfate (DS) as a treatment for patients with AIDS, AIDS related complex (ARC), or asymptomatic HIV infection with or without persistent generalized lymphadenopathy (PGL), and to determine antiviral activity at different doses of DS. Although zidovudine (AZT) has shown promise in prolonging life in patients with AIDS and severe ARC, it has significant blood toxicities. It would be beneficial to combine AZT with another antiviral agent that does not have the same toxicity. DS might be a suitable drug since it has shown antiviral activity against HIV in the laboratory, and in preliminary studies it has shown little toxicity. Also, the combination of DS with AZT has been shown to be more effective than either alone.

DETAILED DESCRIPTION:
Although zidovudine (AZT) has shown promise in prolonging life in patients with AIDS and severe ARC, it has significant blood toxicities. It would be beneficial to combine AZT with another antiviral agent that does not have the same toxicity. DS might be a suitable drug since it has shown antiviral activity against HIV in the laboratory, and in preliminary studies it has shown little toxicity. Also, the combination of DS with AZT has been shown to be more effective than either alone.

The study will begin with 10 patients with AIDS, 10 with ARC, and 10 with asymptomatic HIV infection taking DS by mouth 3 times a day for 24 weeks. If the initial dose of DS is tolerated without significant side effects, the next group of patients will receive a higher dose. A third group of patients will be given either a higher or lower dose depending on the results of the earlier groups. Patients will be evaluated every other week for 12 weeks, then monthly for the remaining 16 weeks. Patients will have the option of continuing DS until the entire study is completed if the drug is well tolerated. Inhaled pentamidine for the prevention of Pneumocystis carinii pneumonia is allowed, but other investigational drugs are not. Drug effects on the HIV virus, immune function, and clinical condition will be monitored during the periodic evaluations.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Aerosolized pentamidine for prophylaxis of Pneumocystis carinii pneumonia (PCP).
* Acetaminophen.
* Ketoconazole.

Consistently positive serum HIV p24 antigen = or > 70 picograms/ml, defined by the Abbott HIV antigen test, on two occasions, each within 1 month prior to entry, separated by at least 72 hours, the last of which must be within 2 weeks of starting therapy. Positive antibody to HIV with a federally licensed ELISA test kit.

Exclusion Criteria

Patients with any negative HIV p24 antigen test within 1 month of entry are excluded. Hemophiliacs are excluded.

Prior Medication:

Excluded within 4 weeks of study entry:

* Biologic response modifiers.
* Zidovudine (AZT) or other antiretroviral agents.
* Other investigational drugs.
* Excluded within 12 weeks of study entry:
* Ribavirin.
* Excluded:
* Ongoing therapy and/or prophylaxis for an AIDS-defining opportunistic infection.
* Anticoagulant drugs.
* Systemic corticosteroids.
* Aspirin.
* Dextran sulfate.
* Sedatives.
* Barbiturates.

Prior Treatment:

Excluded within 2 weeks of study entry:

* Transfusion.

Severe diarrhea:

* = or > 5 loose or watery stools per day. Significant malabsorption:
* > 10 percent weight loss within past 3 months with serum carotene < 75 IU/ml or vitamin A < 75 IU/ml. Transfusion dependent:
* Requiring 2 units of blood > once a month. Active opportunistic infection. Symptomatic visceral Kaposi's sarcoma (KS), progression of KS within 1 month of entry, or concurrent neoplasms other than KS. Basal cell carcinoma of the skin or in situ carcinoma of the cervix. Hemorrhagic diseases such as hemophilia A or B or von Willebrand disease.

Active drug or alcohol abuse sufficient in the investigator's opinion to prevent adequate compliance with study therapy.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60
Dates: Study Completion 1990-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abrams D, Study Chair
Locations (8):
- United States (8):
  - Los Angeles County - USC Med Ctr, Los Angeles, California
  - UCLA CARE Ctr, Los Angeles, California
  - San Francisco AIDS Clinic / San Francisco Gen Hosp, San Francisco, California
  - George Washington Univ Med Ctr, Washington D.C., District of Columbia
  - Univ of Massachusetts Med Ctr, Worcester, Massachusetts
  - Univ of Minnesota, Minneapolis, Minnesota
  - Mem Sloan - Kettering Cancer Ctr, New York, New York
  - Saint Luke's - Roosevelt Hosp Ctr, New York, New York

REFERENCES:
- [Background] Falloon J, et al. 566C80 for the treatment of Pneumocystis carinii pneumonia in AIDS. Int Conf AIDS. 1991 Jun 16-21;7(2):241 (abstract no WB2239)
- [Background] Abrams D, Pettinelli C, Power M, Kubacki VB, Grieco MH, Henry WK. A phase I/II dose ranging trial of oral dextran sulfate in HIV p24 antigen positive individuals (ACTG 060): results of a safety and efficacy trial. Int Conf AIDS. 1989 Jun 4-9;5:404 (abstract no WBP315)